CLINICAL TRIAL: NCT04918940
Title: Post-vaccination Immunization Against SARS-CoV-2 in Patients Undergoing Maintenance With Anti-CD20 Antibodies for Follicular Lymphoma (FL) or Mantle Cell
Brief Title: Efficacy of COVID-19 Vaccination in Patientstreated With Anti-CD20 for Follicular Lymphoma or Mantle Cell Lymphoma
Acronym: VAXIMAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB21.03
Record Dates: First submitted 2021-06-04; First posted 2021-06-09 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Follicular Lymphoma; Mantle Cell Lymphoma
Keywords: Sars-Cov-2 immunization; Vaccination; Rituximab; Obinutuzumab; Maintenance
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-vaccination immunity (Experimental): Samples will be taken after each vaccine injection to perform Sars-Cov-2 serology and Elispot interferon gamma and 3 months after the first vaccine injection
  Interventions: Biological: Determination of COVID-19 vacciantion efficacy

INTERVENTIONS:
Biological: Determination of COVID-19 vacciantion efficacy — Samples will be taken after each vaccine injection to perform Sars-Cov-2 serology and Elispot interferon gamma and 3 months after the first vaccine injection

SUMMARY:
The anti-CD20 monoclonal antibodies, rituximab (R) and obinutuzumab (G), are used as standard maintenance therapy every 2 months for 2 to 3 years in patients with follicular lymphoma (FL) or mantle cell lymphoma (MCL).

This treatment is associated with profound and prolonged B lymphopenia, hypogammaglobulinemia and increased infections. Severe forms of COVID-19 on Rituximab with prolonged carriage of the virus have been reported due to significant impairment of humoral immunity in this context of maintenance therapy.

Therefore, during the COVID-19 epidemic, clinicians are faced with the question of whether to discontinue maintenance therapy or continue treatment. However, the half-life of rituximab is 29 days and lymphopenia continues for up to 9-12 months after stopping injections. Therefore, it is not clear that discontinuation of maintenance therapy will alter the risk of severe SARS-CoV-2.

However, post-vaccination immunization against SARS-CoV-2 by an mRNA vaccine is not known in this context of prolonged treatment with rituximab or obinutuzumab. It is however well established that post-vaccination responses against diphtheria, tetanus, pneumococcus, HBV, or influenza in particular are altered after anti-CD20 antibodies. If the humoral response is crucial in the post-vaccination response, it is also suggested that the preservation of innate immunity and the CD8 response, unaltered by anti-CD20, could also play an important role in the post-vaccination response and virus clearance.

The aim of our study is to evaluate the humoral and post-vaccination T-cell response based on serological data and T-cell production of interferon gamma in response to SARS-CoV-2 specific antigens (Elispot interferon gamma) in this group of patients treated for lymphoma with a long-term anti-CD20 antibody.

ELIGIBILITY:
Inclusion Criteria:

* Age superior to 18 years old
* Patient undergoing maintenance treatment for Mantle Cell Lymphoma or Follicular Lymphoma treated with rituximab or obinutuzumab in complete remission or stable disease between injection #1 and injection #13 or 19 (end of second year or third year)
* Inform consent signed

Exclusion Criteria:

* Documented history of SARS-Cov-2 infection less than 3 months old
* Progressive lymphoma
* Contraindication SARS-Cov-2 vaccination (allergy)
* Refusal of SARS-CoV-2 vaccination
* Patient who has been off rituximab or obinutuzumab therapy for more than 6 months
* Patient not covered by health system
* Pregnant or nursing woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Determination of COVID-19 vaccination immunity | 3 months
  kinetics of anti-SARS-CoV-2 antibody titer
Determination of COVID-19 vaccination immunity | 3 months
  Rate of post-vaccination IFN gamma production

SECONDARY OUTCOMES:
Relapse of lymphoma | one year
  number of relapse of lymphoma
Infections to SARS-Cov-2 | one year
  number of SARS-Cov-2 infection

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Jardin, MD, PhD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No